CLINICAL TRIAL: NCT04581850
Title: Assessment of Sleep Disturbance as a Biomarker of Disease Activity in a Military Population With Posttraumatic Stress Disorder
Acronym: SOMMEPT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PRI01; 2020-A01808-31 (Other: IDRCB)
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTSD patients: This group is composed of patients suffering from an active PTSD
  Interventions: Behavioral: Sleep recording; Behavioral: Cognitive tasks; Other: Questionnaires
- Control group (healthy individuals): This group is composed of healthy individuals.
  Interventions: Behavioral: Sleep recording; Behavioral: Cognitive tasks; Other: Questionnaires

INTERVENTIONS:
Behavioral: Sleep recording — Sleep is recorded at home during 7 nights in a row using a connected headband. The participant also has to fill in a sleep agenda every day.
Behavioral: Cognitive tasks — Working memory and inhibition capacity is assessed during computer-based tasks (2-back and Go/No-Go tasks) at enrollment and 1 month after enrollment.
Other: Questionnaires — The participant has to fill in several questionnaires at enrollment and 1 month after enrollment in order to assess:
  * PTSD severity
  * chronotype
  * Sleep quality
  * Daytime sleepiness
  * Mood state
  * Depression
  * Mental disorders and their consequences

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) is a public health problem due to both its chronic nature and the low response rate to conventional therapies.

Sleep disorders are the first cause of complaint in patients with PTSD due to night awakenings, difficulty to fall asleep and nightmares.

According to a part of the scientific community, replicative traumatic nightmares represent PTSD's basis mechanism. Traumatic nightmares generate disabling symptoms such as anxiety reactions, while maintaining the symptoms by depriving the individual of good quality sleep. Traumatic nightmares may thus be a sign of PTSD seriousness and chronicity, although their physiological basis remain poorly known.

In the military population, which is highly exposed to psychological traumatism, PTSD prevalence is very high and is associated with severe intensity patterns, a very high frequency of replicative nightmares and a low response to conventional therapies.

ELIGIBILITY:
Inclusion Criteria:

* Military or former military
* Age between 18 and 65 years old
* PTSD group : with a PTSD diagnosis
* Control group : without any sleep, psychiatric or neurologic pathology

Exclusion Criteria:

* Diagnosis of progressive psychiatric pathology prior to the traumatic event responsible for PTSD
* Sleep pathology prior to the traumatic event responsible for PTSD
* Neurological pathology or severe head injury within the last 3 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of patients suffering from an active PTSD and healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a Sleep Efficiency Index (SEI) < 80%. | 1 month after enrollment
  The sleep efficiency index (SEI) is defined by the ratio TST/TIB with TST being Total Sleep Time and TIB being Time In Bed.
  TST and TIB will be assessed objectively, at home, using a connected headband (DREEM®, Rythm Paris).
  A Sleep Efficiency Index (SEI) < 80% is considered to be a poor quality, low-efficiency night.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hôpoital d'Instruction des Armées Percy, Clamart
  - 52e Antenne Médicale, Mailly-le-Camp
  - Hôpital d'Instruction des Armées Laveran, Marseille
  - 29e Antenne Médicale, Mourmelon-le-Grand
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saguin E, Feingold D, Sipahimalani G, Quiquempoix M, Roseau JB, Remadi M, Annette S, Guillard M, Van Beers P, Lahutte B, Leger D, Gomez-Merino D, Chennaoui M. PTSD Symptom Severity Associated With Sleep Disturbances in Military Personnel: Evidence From a Prospective Controlled Study With Ecological Recordings. Depress Anxiety. 2025 Apr 25;2025:8011375. doi: 10.1155/da/8011375. eCollection 2025. PMID 40370761